CLINICAL TRIAL: NCT05740124
Title: Workplace Fall Prevention Through Slip Recovery Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Michael Madigan, Professor, Virginia Polytechnic Institute and State University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-853
Record Dates: First submitted 2023-01-21; First posted 2023-02-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Accidental Fall
Keywords: slips; balance recovery; perturbation-based balance training; balance training; falls

STUDY DESIGN:
Intervention Model Description: We selected N/A for study phase because this study involves a behavioral intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Slip recovery training (Experimental): Once weekly sessions of slip recovery training for 3 or 6 weeks. Each session will be 20 minutes of training. Training will involve volitional and reactive stepping movements that mimic the movements necessary to recover balance after slipping while walking.
  Interventions: Behavioral: slip recovery training
- Alternative balance training (Active Comparator): Once weekly sessions of balance training for 3 or 6 weeks. Each session will be 20 minutes of training. Training will involve standing balance under varied sensory conditions, and tandem walking forward and backward under varied sensory conditions.
  Interventions: Behavioral: alternative balance training

INTERVENTIONS:
Behavioral: slip recovery training — Participants practice volitional and reactive stepping responses that mimic those needed when recovering balance after slipping.
  Arms: Slip recovery training
Behavioral: alternative balance training — Participants practice standing and walking under varied sensory conditions.
  Arms: Alternative balance training

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of applying slip recovery training, a novel balance training exercise intervention, to workers who are at increased risk of slip-induced falls. This will be done via field studies with industrial partners. Note that the slip recovery training is not a device or drug. It is a detailed exercise regimen that aims to improve the the ability to recover balance after slipping.

The main specific aims are are:

* To investigate the feasibility of on-site slip recovery training
* To validate field assessments for evaluating slip recovery training efficacy in subsequent research

Participants will complete 3-6 once-weekly sessions of slip recovery training, answer daily text messages indicating any falls they experience while working over the 12 weeks after completing slip recovery training, and a subset of workers will be asked to participate in focus group discussions after the 12 weeks to provide information on the long-term feasibility of slip recovery training. A group of workers at Virginia Tech will also be asked to complete a laboratory session of testing during which they will be exposed to a laboratory-induced slip so that gold-standard measures of slip-induced fall recovery can be used to validate field assessments.

Workers who complete slip recovery training will be compared to another group of workers who complete an alternative balance training that should improve balance but not improve slip recovery that is targeted by slip recovery training.

ELIGIBILITY:
Inclusion Criteria:

* Virginia Tech workers in Dining Services, Facilities and Housekeeping, and construction.
* Veolia field workers in water distribution and water main construction
* age 18-65 years old
* willing to complete 3 or 6 training sessions, lab testing session, and daily falls tracking for 12 weeks

Exclusion Criteria:

* weigh over 250 pounds
* answer 'no' to all questions of the Physical Activity Readiness Questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
evaluation of recruitment methods | 2 years
  number of prospective participants who contact the investigators with interest in participating
evaluation of screening methods | 2 years
  percentage of prospective participants who are deemed a poor fit for the study based upon not passing the Physical Activity Readiness Questionnaire.
worker adherence to slip recovery training | during 3 or 6 weeks of balance training
  average number of slip recovery training sessions completed across all participants assigned to slip recovery training
worker adherence to alternative balance training | during 3 or 6 weeks of balance training
  average number of alternative balance training sessions completed across all participants assigned to alternative balance training
worker retention during 12 weeks of falls tracking | during the12 weeks after completing the training intervention
  average number of weeks participants responded to text messages from investigators regarding slips and falls
lab-induced slip outcome (fall or recovery) | during the laboratory testing session that will take place within one week of completing training intervention
  a binary measure determined based on the force applied to the safety harness worn by all participants when exposed to a laboratory-induced slip
lab-induced slip distance | during the laboratory testing session that will take place within one week of completing training intervention
  the distance the slipping foot slides when exposed to a laboratory-induced slip
lab-induced slip peak slip speed | during the laboratory testing session that will take place within one week of completing training intervention
  the peak speed of the slipping foot during slip when exposed to a laboratory-induced slip
efficacy of field assessments of balance | during the field session one week after completing the training intervention
  Pearson product correlation coefficient between field assessment of slip distance and lab-induced slip distance

SECONDARY OUTCOMES:
field assessment of slip distance | one week after intervention
  the distance the slipping foot slides when exposed to a slip induced in the field
field assessment of slip distance | 12 weeks after intervention
  the distance the slipping foot slides when exposed to a slip induced in the field
field assessment of peak slip speed | one week after intervention
  the maximum slipping speed of the foot during recovery from an induced slip
field assessment of peak slip speed | 12 weeks after intervention
  the maximum slipping speed of the foot during recovery from an induced slip
postural sway during quiet standing | one week after intervention
  mean center of pressure speed
postural sway during quiet standing | 12 weeks after intervention
  mean center of pressure speed
dynamic balance performance | one week after intervention
  maximum number of consecutive backward toe-to-heel steps completed while walking three times along a 3cm-wide, 3m-long beam on the floor without touching the ground
dynamic balance performance | 12 weeks after intervention
  maximum number of consecutive backward toe-to-heel steps completed while walking three times along a 3cm-wide, 3m-long beam on the floor without touching the ground
number of falls while working during 12-week follow up | during the 12 week follow up after intervention
  determined using a daily text message questionnaire
number of near-falls while working during 12-week follow up | during the 12 week follow up after intervention
  determined using a daily text message questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Madigan, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No